CLINICAL TRIAL: NCT05268731
Title: Defining the Clinical Success of Different Percutaneous Transhepatic Biliary Drainage Procedures
Brief Title: Clinical Success of Different Percutaneous Transhepatic Biliary Drainage Procedures
Acronym: TransHepatic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: Helios Kliniken Schwerin (Other)
Responsible Party: Sponsor
Other Study IDs: PTBD retro 003
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Extrahepatic Cholestasis
Keywords: Extrahepatic Cholestasis; Self Expandable Metallic Stents; Drainage
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extrahepatic bile duct obstruction and failed ERCP: Patients with extrahepatic bile duct obstruction and obstructive jaundice have received a percutaneous transhepatic biliary drainage.
  The choice between an insertion of an external or an external/internal drainage has been made during the procedure depending on whether the guide wire could be accessed to the jejunum/duodenum or not.
  The choice between internal/external drainage or a primary metal stent has been made by the investigators preference or was made on the basis of an existing malign bile duct obstruction or not.
  Interventions: Procedure: External plastic endoprosthesis; Procedure: Combined external internal plastic endoprosthesis; Procedure: Primary metal stent

INTERVENTIONS:
Procedure: External plastic endoprosthesis — Ultrasound- or fluoroscopy-guided bile duct puncture with insertion of an external plastic endoprosthesis if the duodenum or jejunum cannot be accessed by a guide wire
Procedure: Combined external internal plastic endoprosthesis — Ultrasound- or fluoroscopy-guided bile duct puncture with insertion of an external/internal plastic endoprosthesis if the duodenum or jejunum can be accessed by a guide wire. No definitive drainage intended in initial procedure.
Procedure: Primary metal stent — Ultrasound- or fluoroscopy-guided bile duct puncture with insertion of a self-expanding metal stent if the duodenum or jejunum can be accessed by a guide wire. A definitive drainage is intended in the initial procedure, for example in patients with malign bile duct obstruction

SUMMARY:
The clinical success of percutaneous transhepatic biliary drainage procedures (PTBDs) is usually measured by the the decrease of the serum bilirubin value. However, the bilirubin value can be biased by other disease conditions. Furthermore, the time course of the decrease of the bilirubin value after technically successful PTBD is not well known. Serum gamma-glutamyl transferase (GGT), a liver enzyme which is typically elevated in cholestatic liver diseases, might be a good alternative to bilirubin as an indicator for the clinical success of PTBDs. The aim of this study is to analyse the bilirubin level and the GGT level in patients with technically successful PTBD.

DETAILED DESCRIPTION:
The medical records of adult patients who have received a technically successful PTBD will be screened sytematically in terms of bilirubin and GGT values in the follow up of 4 weeks after the intervention. Bilirubin and GGT values have been routinely examinated every 1 to 3 days. PTBD comprises external plastic endoprosthesis, combined external and internal endoprosthesis and primary metal stent insertion. The respective three procedures are considered separately. As PTBD is a rare intervention which is used after failed or impossible endoscopic retrograde cholangiopancreaticography (ERCP) medical records will be screened from 2002 to 2022 (20 years). It is expected that for example a decrease of GGT after three days might indicate a successful procedure. This in turn might has an impact on the early demission of the patient. On the other side, the precise definition of successful PTBD by bilirubin or GGT value might help to make this procedure better comparable to other alternative biliary drainage procedures such as endoscopic ultrasound-guided biliary drainage.

ELIGIBILITY:
Inclusion Criteria:

* technically successful PTBD

Exclusion Criteria:

* technically not successful PTBD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extrahepatic bile duct obstruction and failed or impossible ERCP
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Bilirubin value | 4 weeks
  Change of serum bilirubin value
GGT value | 4 weeks
  Change of serum bilirubin value

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, MD, Principal Investigator — Theresienkrankenhaus Mannheim, University of Heidelberg
Locations (1):
- Helios Kliniken Schwerin, Schwerin, Germany

IPD SHARING:
Plan to Share IPD: No
All data of the study will be available on request

REFERENCES:
- [Result] Born P, Rosch T, Triptrap A, Frimberger E, Allescher HD, Ott R, Weigert N, Lorenz R, Classen M. Long-term results of percutaneous transhepatic biliary drainage for benign and malignant bile duct strictures. Scand J Gastroenterol. 1998 May;33(5):544-9. doi: 10.1080/00365529850172142. PMID 9648997
- [Result] Tsai CC, Mo LR, Lin RC, Kuo JY, Chang KK, Yeh YH, Yang SC, Yueh SK, Tsai HM, Yu CY. Self-expandable metallic stents in the management of malignant biliary obstruction. J Formos Med Assoc. 1996 Apr;95(4):298-302. PMID 8935298